CLINICAL TRIAL: NCT04398121
Title: Narrow Band Imaging in Oral Cavity Cancer-defining the Tumour Border
Brief Title: NBI in Oral Cavity Cancer
Status: Completed | Type: Observational
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Other Study IDs: 273124
Record Dates: First submitted 2020-05-19; First posted 2020-05-21 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Oral Cancer
Keywords: tumour border; tumor margin; narrow band imaging; oral cancer; oral carcinoma
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Oral cancer starts in the mucosa of the mouth and the most common site is the tongue and gingiva. One of the most important issues for the prognosis is to surgically remove all the cancer, at the sides as well as at the deep margin. To accomplish that, it is crucial to identify the border between tumour and healthy tissue. Traditionally white light from a head light or operation theatre lamp is used to illuminate the area of the tumour. Narrow Band Imaging (NBI) is an optical technique where ordinary white light is filtered so only the blue light in it is used. Illuminating the mucosa with this blue light through an endoscope with high definition image, makes the blood vessels appear more clearly. The altered blood vessels that the cancer produce can thereby be seen and mark the area where the tumour starts.

This study examines if NBI is helpful in the decision of where the border between the cancer and the normal mucosa is. If so, NBI might improve the possibility to remove all cancer tissue compared to using the ordinary white light.

This study will also increase the knowledge about the NBI technique, which is helpful in the examination of patients with suspected head and neck cancers and at the follow-up of patients after treatment.

Participants are patients with oral cancer presenting at the otorhinolaryngology department in Örebro University hospital in Sweden for surgical treatment. The surgery will be done in the usual fashion but the mucosa surrounding the tumour will also be illuminated by NBI and this picture of the vessels will be compared to the microscopic analysis by the pathologist, the so called PAD. Thereby we seek to compare the border in white light to the border seen with NBI.

DETAILED DESCRIPTION:
Patients with primary oral cavity cancer will be examined with Narrow Band Imaging (NBI) at the time of surgery. Olympus® equipment will be used together with straight 5,9 mm endoscopes.

First the tumour border seen in white light will be defined. Thereafter endoscopic examination with white light and NBI will be performed and recorded. Then the tumour border seen in white light will be marked with dots by monopolar diathermy. Finally the area is examined again with NBI and if the tumour border is seen outside the border seen in white light, that area is marked by a suture for the pathology report.

Since the purpose of this study is to gain knowledge of NBI in oral cavity cancer, the resection margin will be marked at least 10mm from the tumour border as it is seen in white light in the ordinary fashion. However there are evolving evidence that NBI better delineate tumour border in larynx and some data for the oral cavity, therefore any suspected mucosa according to NBI outside the ordinary resection margin will be included with a small margin.

There is no uniform definition of the NBI pattern in oral cavity cancer. The planned criteria is changed IPCL type III/IV according to Takano (see ref.) and so called "marked brown dots" as criteria for precancerous or cancerous mucosa according to NBI.

The tumour border in white light and NBI will be compared and PAD is considered gold standard.

To reach 80% power with 5 % type 1 error, two-sided test, and 25% of the examinations anticipated to show different tumour border with NBI, 49 participants will be needed.

ELIGIBILITY:
Inclusion Criteria:

Biopsy proven squamous cell carcinomaI. International Statistical Classification of Diseases and Related Health Problems (ICD) 10 C02-C06.

Exclusion Criteria:

* former extensive surgery in the oral cavity that effects the examination
* former radiation to the oral cavity
* patients not suitable for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be patients with oral cancer presenting for treatment at our clinic. All patients that meet the eligibility criteria will be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
NBI tumour border | 4 weeks
  the possibility to determine the tumour border in the mucosa with NBI compared to white light.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Knutsson, Assoc. Prof., Principal Investigator — Region Örebro County
Locations (1):
- Örebro University Hospital, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymised data of the NBI-picture in relation to PAD will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication
Access Criteria: Coded, computerized IPD will be available upon a request with the serious intention to improve the scientific knowledge and transparency.

REFERENCES:
- [Background] Takano JH, Yakushiji T, Kamiyama I, Nomura T, Katakura A, Takano N, Shibahara T. Detecting early oral cancer: narrowband imaging system observation of the oral mucosa microvasculature. Int J Oral Maxillofac Surg. 2010 Mar;39(3):208-13. doi: 10.1016/j.ijom.2010.01.007. Epub 2010 Feb 24. PMID 20185271
- [Background] Ni XG, He S, Xu ZG, Lu N, Gao L, Yuan Z, Zhang YM, Lai SQ, Yi JL, Wang XL, Zhang L, Li XY, Wang GQ. [Application of narrow band imaging endoscopy in the diagnosis of laryngeal cancer]. Zhonghua Er Bi Yan Hou Tou Jing Wai Ke Za Zhi. 2010 Feb;45(2):143-7. Chinese. PMID 20398512
- [Background] Piazza C, Del Bon F, Paderno A, Grazioli P, Perotti P, Barbieri D, Majorana A, Bardellini E, Peretti G, Nicolai P. The diagnostic value of narrow band imaging in different oral and oropharyngeal subsites. Eur Arch Otorhinolaryngol. 2016 Oct;273(10):3347-53. doi: 10.1007/s00405-016-3925-5. Epub 2016 Feb 15. PMID 26879990
- [Background] Farah CS. Narrow Band Imaging-guided resection of oral cavity cancer decreases local recurrence and increases survival. Oral Dis. 2018 Mar;24(1-2):89-97. doi: 10.1111/odi.12745. PMID 29480612
- [Background] Tirelli G, Piovesana M, Marcuzzo AV, Gatto A, Biasotto M, Bussani R, Zandona L, Giudici F, Boscolo Nata F. Tailored resections in oral and oropharyngeal cancer using narrow band imaging. Am J Otolaryngol. 2018 Mar-Apr;39(2):197-203. doi: 10.1016/j.amjoto.2017.11.004. Epub 2017 Nov 10. PMID 29150027